CLINICAL TRIAL: NCT06276166
Title: Study of the Joint Trajectory of Frailty and Cognitive Dysfunction Among Community-dwelling Older Adults
Brief Title: Trajectory of Frailty and Cognitive Dysfunction in Older Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Zheng Li (Other)
Responsible Party: Sponsor-Investigator, Zheng Li, Professor, Peking Union Medical College
Organization: Peking Union Medical College (Other)
Other Study IDs: 72374215
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Frailty; Cognitive Dysfunction; Community-dwelling Older Adults
MeSH Terms: conditions — Frailty; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood glucose, Blood lipid, Glycosylated hemoglobin, Homocysteine, C-reactive protein, Interleukin
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults: Older adults without clear diagnosis of any type of dementia, neurological diseases, and mental disorders that affecting cognitive function.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
To explore the heterogeneity of the development trend of frailty and cognitive function of older adults.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, the older adults will be selected from community health service centers in four districts of Beijing. Frailty and cognitive function of the older adults will be assessed for a 24-month longitudinal multi-time (baseline, 6, 12 and 24 months). The heterogeneity of the development trend of frailty and cognitive function will be explored, and the subgroups of joint development trajectory of frailty and cognitive impairment will be classified, so as to identify high-risk populations that need to be managed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years.
* Older adults with clear consciousness, ability of simple written and verbal communication.
* They volunteered to participate in this study, and signed an informed consent.

Exclusion Criteria:

* A clear diagnosis of any type of dementia.
* There are neurological diseases that clearly lead to cognitive dysfunction, such as severe cerebrovascular disease, brain trauma, intracranial tumors, etc.
* They have been clearly diagnosed with mental disorders affecting cognitive function, including schizophrenia, depression, bipolar disorder, etc.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults without clear diagnosis of any type of dementia, neurological diseases, and mental disorders that affecting cognitive function.
Sampling Method: Non-Probability Sample
Enrollment: 934 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Frailty | Baseline, 6 month, 12 month, and 24 month
  Frailty was evaluated by the Fried phenotype model, which was proposed and validated by Fried and colleagues, and is the most widely adopted model, generally regarded as the standard model for physical frailty. In Fried's model, the frailty phenotype is based on the following five components: slowness (gait speed), weakness (hand grip), weight loss, exhaustion, and low physical activity.
Cognitive function | Baseline, 6 month, 12 month, and 24 month
  The method to assess objective cognitive function is Montreal Cognitive Assessment-Beijing version for Chinese, which is a classical tool to screen for MCI, including 7 cognitive domains (visuospatial and executive function, naming, attention, language, abstraction, delayed recall, and orientation). The total score of the scale is 30, with higher scores indicating better cognitive function. The Mini-Mental State Examination (MMSE) which included 30 questions to measure the cognitive status will be also performed to assess objective cognitive function.
  In addition, We use the 9-items subjective cognitive decline questionnaire (SCD-Q9) to measure the symptoms of subjective cognition. The SCD-Q9 is a simple and quick screening scale to identify those who suffer from MCI from general populations. SCD-Q9 lists the 9 core items of SCD symptoms and contains 2 dimensions and 9 items.

OTHER OUTCOMES:
Health status and life style | Baseline, 6 month, 12 month, and 24 month
  Data on health status (disease, hearing) and lifestyle (diet, sleep, exercise) of the elderly were obtained through self-made questionnaires.
Activities of daily life (ADLs) | Baseline, 6 month, 12 month, and 24 month
  The Chinese version of the ADLs scale revised by Zhang will be utilized to identify the ability to perform the activities. A summary score for each item ranges from 1 (require no help) to 4 (unable to do it at all) points. The first eight items measure Basic Activities of Daily Living (BADLs), with a total score of 8~32. The last 12 items are about Instrumental Activities of Daily Living (IADLs), with a total score of 12~48. The lower the score, the lower the degree of dependence on daily life.
Anxiety | Baseline, 6 month, 12 month, and 24 month
  General anxiety disorder-7 (GAD-7) will be utilized, which is a seven-question screening tool that identifies whether a complete assessment for anxiety is indicated. Scoring Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Apathy | Baseline, 6 month, 12 month, and 24 month
  The apathy subscale (GDS-3A) of the GDS-15 consists of the following three items (score range 0-3 points) will be utilized: (i) Have you dropped many of your activities and interests?; (ii) Do you prefer to stay at home, rather than going out and doing new things?; and (iii) Do you feel full of energy?.
Perceived social support | Baseline, 6 month, 12 month, and 24 month
  The perceived social support scale (PSSS) consists of 12 items, which are divided into three dimensions: family support, friends support and other support. The scale was developed by Zimet et al. and has a favourable internal consistency (Cronbach's α = 0.85-0.91). Each item is scored from 1 (strongly disagree) to 7 (strongly agree), and the total score ranges from 7 to 84. The higher the score is, the higher the level of social support the individual feels.
Social network | Baseline, 6 month, 12 month, and 24 month
  Lubben Social Network Scale (LSNS-6) includes a set of three items on family and a comparable set of three items on friends, asking about frequency of contact and emotional closeness. More specifically, the items address the number of network members whom the respondent (a) sees or hears from at least once a month, (b) feels at ease talking about private matters, and (c) feels close enough to call for help. The respondent answered each question by selecting a value on a 6-point scale (ranging from 0 = none to 5 = nine or more). Each family/friend subscale could range from 0 to 15, and the total score from 0 to 30. Higher scores indicate stronger ties with family or friends.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Li, Study Chair — Chinese Academy of Medical Sciences & Peking Union Medical College